CLINICAL TRIAL: NCT07117864
Title: Exploration of the Safety and Efficacy of T-DXd Concurrent With Brain Radiotherapy in Patients With Brain Metastases HER2-positive/HER2-low Advanced Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: QIAO LI (Other)
Responsible Party: Sponsor-Investigator, QIAO LI, Director, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/376-4656; NCC4774 (Registry Identifier: T-DXd concurrent with brain radiotherapy in patients with brain metastases HER2-positive/HER2-low ABC)
Record Dates: First submitted 2025-07-09; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T-DXd concurrent brain radiotherapy (Experimental): T-DXd：5.4mg/kg ivgtt Q3w SRT/WBRT
  Interventions: Combination Product: T-DXd concurrent brain radiotherapy

INTERVENTIONS:
Combination Product: T-DXd concurrent brain radiotherapy — T-DXd：5.4mg/kg ivgtt Q3w SRT/WBRT

SUMMARY:
A study on the safety and efficacy of T-DXd in combination with local radiotherapy for brain metastases in HER2-Positive and HER2-Low breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 and ≤75 years with histologically confirmed breast cancer.
2. ECOG performance status of 0 to 2.
3. HER2-positive or HER2-low invasive breast cancer, defined as:

   HER2-positive: IHC 3+ or IHC 2+ with FISH amplification; HER2-low: IHC 2+ without FISH amplification, or IHC 1+.
4. Confirmed diagnosis of breast cancer brain metastases.
5. Patients may have received prior chemotherapy (from first-line to multiple lines), HER2-targeted therapy (monoclonal antibodies), endocrine therapy, and immunotherapy.
6. Adequate organ function as defined below:

   Hematology:

   Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelet count (PLT) ≥ 80 × 10⁹/L (no blood transfusion within 14 days prior to first dose); Hemoglobin (Hb) ≥ 80 g/L;

   Serum biochemistry:

   Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); ALT and AST ≤ 2.5 × ULN; Blood urea nitrogen (BUN) and serum creatinine ≤ 1.5 × ULN;

   Cardiac function:

   Echocardiography: Left ventricular ejection fraction (LVEF) ≥ 45%.
7. Subjects must voluntarily participate in the study and provide signed informed consent.

Exclusion Criteria:

1. Tumor-Related Symptoms and Treatments

   1. Uncontrolled moderate to large pleural effusion, ascites, or pericardial effusion requiring repeated drainage;
   2. Imaging (CT or MRI) showing tumor invasion of major blood vessels, or cases deemed by the investigator as highly likely to cause fatal hemorrhage due to vascular invasion during the study period;
   3. Signs of meningeal irritation such as neck stiffness, seizures, or cognitive impairment, or confirmed leptomeningeal metastasis by imaging (CT or MRI) or lumbar puncture;
   4. Uncontrolled or symptomatic hypercalcemia (defined as ionized calcium > 1.5 mmol/L, serum calcium > 12 mg/dL, or albumin-corrected serum calcium > ULN), or symptomatic hypercalcemia requiring continued bisphosphonate treatment;
   5. Prior cranial radiotherapy;
   6. Prior treatment with trastuzumab deruxtecan (T-DXd).
2. Comorbidities / Medical History

   1. History of other malignancies for which the patient received any systemic anti-cancer therapy or local treatment (including surgery or radiotherapy), except for adequately treated cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin;
   2. Major surgery unrelated to breast cancer within 4 weeks prior to enrollment, or incomplete recovery from such surgery (diagnostic biopsies and PICC line placement are permitted);
   3. Known or suspected autoimmune diseases, except for the following conditions:

      Hypothyroidism due to autoimmune thyroiditis managed with hormone replacement therapy; Stable Type I diabetes mellitus with controlled blood glucose;
   4. Presence of interstitial lung disease (ILD), non-infectious pneumonitis, or uncontrolled systemic diseases (e.g., diabetes, pulmonary fibrosis, acute pneumonia);
   5. HIV infection or known AIDS; active hepatitis (HBV defined as HBV-DNA ≥ 500 IU/mL; HCV defined as HCV-RNA above the lower limit of detection); concurrent HBV and HCV infection; autoimmune hepatitis;
   6. Severe infections within 4 weeks before first dose (e.g., bacteremia or severe pneumonia requiring hospitalization), or active infections requiring systemic antibiotic therapy of CTCAE grade ≥2 within 2 weeks before first dose, or unexplained fever >38.5°C during screening or prior to first dose (fever deemed tumor-related may be eligible at the investigator's discretion); evidence of active tuberculosis within 1 year prior to first dose;
   7. Previous or planned allogeneic bone marrow transplantation or solid organ transplantation;

   Severe or uncontrolled cardiovascular disease, including but not limited to:

   History of heart failure or systolic dysfunction (LVEF < 45%); High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate > 100 bpm, significant ventricular arrhythmias (e.g., ventricular tachycardia), or high-grade atrioventricular (AV) block (e.g., Mobitz type II second-degree or third-degree AV block); Angina requiring anti-anginal medications; Clinically significant valvular heart disease; Transmural myocardial infarction on ECG; Poorly controlled hypertension (systolic BP >180 mmHg and/or diastolic BP >100 mmHg);
3. Known hypersensitivity to the investigational drug or any of its excipients, or a history of severe hypersensitivity reactions to other monoclonal antibodies.
4. Pregnant or breastfeeding women, women of childbearing potential with a positive baseline pregnancy test, or women of childbearing potential unwilling to use effective contraception during the study.
5. History of confirmed neurological or psychiatric disorders, including epilepsy or dementia; known history of psychiatric medication abuse, alcoholism, or substance abuse.
6. Any other condition that, in the investigator's judgment, makes the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
brain progression-free survival | At the end of Cycle 1(each cycle is 21 days)
  brain progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Li, MD, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China